CLINICAL TRIAL: NCT03472846
Title: MicroRNAs Levels in Women With Postmenopausal Osteoporosis Under Antiresorptive or Osteoanabolic Treatment
Brief Title: MiDeTe - microRNA Levels Under Denosumab and Teriparatide Therapy in Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: St. Vincent Hospital, Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christian Muschitz, OA Priv. Doz. Dr. Christian Muschitz, Medical University of Vienna
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MIDETE
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Postmenopausal Osteoporosis; Diabetes Type 2
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Diabetes Mellitus, Type 2 | interventions — Denosumab; Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 - DMAB (Active Comparator): postmenopausal women without type 2 diabetes mellitus treated with denosumab
  Interventions: Drug: Prolia, 60 Mg/mL Subcutaneous Solution
- Group 2 - TPTD (Active Comparator): postmenopausal women with type 2 Diabetes mellitus treated with teriparatide
  Interventions: Drug: Teriparatide
- Group 3 - DMAB (Active Comparator): postmenopausal women with type 2 diabetes mellitus treated with denosumab
  Interventions: Drug: Prolia, 60 Mg/mL Subcutaneous Solution
- Group 4 - TPTD (Active Comparator): postmenopausal women without type 2 diabetes mellitus treated with teriparatid
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Prolia, 60 Mg/mL Subcutaneous Solution — antiresorptive treatment with Prolia
  Arms: Group 1 - DMAB; Group 3 - DMAB
Drug: Teriparatide — osteoanabolic treatment with Forsteo
  Arms: Group 2 - TPTD; Group 4 - TPTD

SUMMARY:
The aim of this study is the quantitative determination of bone-specific microRNAs in the serum of postmenopausal women with osteoporosis during antiresorptive or osteoanabolic therapy.

DETAILED DESCRIPTION:
Primarily the influence of the therapeutic treatment on the microRNA concentration in the serum (treatment-response) and the relation between microRNA serum levels and changes of the bone mineral density will be investigated.

These data will help to examine the use of microRNAs as novel diagnostic biomarkers for the diagnosis of osteoporosis and targeted therapeutic treatment of patients.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Age 60-80 years
* T-score according to DXA: <-2.5
* indication for osteoporosis therapy according to international guidelines

Exclusion Criteria:

* Diabetes mellitus type 1
* renal insufficiency III-V °
* Cirrhosis hepatis (Child B or higher)
* Chronic alcohol abuse
* rheumatic disease (RA, SpA, SLE)
* Malignancies (<5 years)
* Eating Disorder (anorexia nervosa, bulimia)
* bone-specific pretreatment (DMAB, TPTD, strontium ranelate, SERMs) Bisphosphonate treatment is allowed

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
detection of microRNA concentration in serum | 24 months
  influence of antiresorptive or osteoanabolic Treatment on microRNA levels in postmenopausal women with osteoporosis

SECONDARY OUTCOMES:
microRNAs and changes in bone metabolism under treatment | 24 months
  correlation of microRNA with bone turnover markers, fracture risk, BMD

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna; St. Vincent Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided